CLINICAL TRIAL: NCT01372150
Title: A MULTICENTER, RANDOMIZED, DOUBLE-BLIND, PLACEBO-CONTROLLED, FLUOXETINE-REFERENCED, PARALLEL-GROUP STUDY TO EVALUATE THE EFFICACY, SAFETY AND TOLERABILITY OF DESVENLAFAXINE SUCCINATE SUSTAINED RELEASE (DVS SR) IN THE TREATMENT OF CHILDREN AND ADOLESCENT OUTPATIENTS WITH MAJOR DEPRESSIVE DISORDER
Brief Title: A Study Of DVS SR In Treatment Of Children And Adolescent Outpatients With MDD
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: B2061014; 3151A6-3356 (Other: Alias Study Number); 2008-002063-13 (EudraCT Number)
Record Dates: First submitted 2011-06-09; First posted 2011-06-13 (Estimated); Results first posted 2015-11-20 (Estimated); Last update posted 2019-01-15 (Actual); Status verified 2019-01

CONDITIONS: Major Depressive Disorder
Keywords: major depressive disorder; MDD; depression
MeSH Terms: conditions — Depressive Disorder, Major; Depression | interventions — Fluoxetine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- DVS SR (Experimental)
  Interventions: Drug: desvenlafaxine succinate sustained release
- Fluoxetine (Other): Active control for assay sensitivity
  Interventions: Drug: fluoxetine
- Placebo (Experimental)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: desvenlafaxine succinate sustained release — Subjects randomized to DVS SR group receive 25, 35 or 50 mg/day based on subject weight at the Baseline visit. DVS SR provided as oral tablets.
  Arms: DVS SR
Drug: fluoxetine — Subjects randomized to the fluoxetine group receive 20 mg/day. Fluoxetine provided as oral capsules
  Arms: Fluoxetine
Drug: placebo — Subjects randomized to the placebo group receive corresponding placebo tablets and/capsules
  Arms: Placebo

SUMMARY:
This is a Double-blind Study Evaluating Desvenlafaxine Succinate (DVS SR) Sustained Release vs Placebo in the Treatment of Children and Adolescent Outpatients with Major Depressive Disorder (MDD).

ELIGIBILITY:
Inclusion Criteria:

* Age >=7 and <18 years of age
* Primary diagnosis of major depressive disorder (MDD)
* CDRS-R score >40

Exclusion Criteria:

* History of suicidal behaviour, or requires precaution against suicide
* Not in generally healthy medical condition
* History of psychosis or bipolar disorder
* Seizure disorder

Ages: 7 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 340 (Actual)
Dates: Start 2011-11-17 (Actual); Primary Completion 2015-03-20 (Actual); Study Completion 2015-03-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (43):
- United States (41):
  - Harmonex Neuroscience Research, Inc., Dothan, Alabama
  - Dedicated Clinical Research, Goodyear, Arizona
  - University of Arizona Clinical and Translational Science Center (CATS), Tucson, Arizona
  - University of Arizona College of Medicine Dept of Psychiatry, Tucson, Arizona
  - Arkansas Psychiatric Clinic Clinical Research Trials, P.A., Little Rock, Arkansas
  - ATP Clinical Research, Inc. 1, Costa Mesa, California
  - Behavioral Research Specialists, LLC, Glendale, California
  - Synergy Clinical Research Center, National City, California
  - Neuropsychiatric Research Center of Orange County, Orange, California
  - Pacific Clinical Research Medical Group, Orange, California
  - Sharp Mesa Vista Hospital, San Diego, California
  - Elite Clinical Trials, Incorporated, Wildomar, California
  - Children's Hospital Colorado, Aurora, Colorado
  - Amedica Research Institute, Incorporated, Hialeah, Florida
  - Clinical Neuroscience Solutions, Inc., Orlando, Florida
  - Kolin Research Group, Winter Park, Florida
  - Winter Park Memorial Hospital, Winter Park, Florida
  - Atlanta Center for Medical Research, Atlanta, Georgia
  - Institute for Behavioral Medicine, Smyrna, Georgia
  - Psychiatric Associates, Overland Park, Kansas
  - Lake Charles Clinical Trials,, Lake Charles, Louisiana
  - Neuroscientific Insights, Rockville, Maryland
  - Precise Research Centers, Flowood, Mississippi
  - Midwest Research Group, Saint Charles, Missouri
  - St. Charles Psychiatric Associates - Midwest Research Group, Saint Charles, Missouri
  - Heartland Pharma Developments, North Platte, Nebraska
  - Creighton University, Omaha, Nebraska
  - Center for Psychiatry and Behavioral Medicine, Incorporated, Las Vegas, Nevada
  - Cincinnati Children's Hospital Medical Center (New), Cincinnati, Ohio
  - Nina F. Wimpie, MD Pediatrics, Middleburg Heights, Ohio
  - North Star Medical Research, LLC, Middleburg Heights, Ohio
  - IPS Research Company, Oklahoma City, Oklahoma
  - Cutting Edge Research Group, Oklahoma City, Oklahoma
  - Paradigm Research Professionals, LLC, Oklahoma City, Oklahoma
  - Summit Research Network (Oregon), Incorporated, Portland, Oregon
  - Clinical Neuroscience Solutions, Inc, Memphis, Tennessee
  - Focus & Balance, LLC, San Antonio, Texas
  - Grayline Clinical Drug Trials, Wichita Falls, Texas
  - Northwest Clinical Research Center, Bellevue, Washington
  - Summit Research Network (Seattle) LLC, Seattle, Washington
  - Rogers Center For Research And Training, Milwaukee, Wisconsin
- Mexico (2):
  - Hospital Aranda de la Parra S.A. de C.V., León, Guanajuato
  - CIT - Neuropsique, S.C., Monterrey, Nuevo León

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B2061014&StudyName=A%20Study%20Of%20DVS%20SR%20In%20Treatment%20Of%20Children%20And%20Adolescent%20Outpatients%20With%20MDD

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Placebo tablets and capsules administered once daily for 8 weeks (treatment phase), followed by placebo tablets and capsules administered once daily as appropriate for 1 week (taper/transition phase).
- Fluoxetine: Fluoxetine capsules 10 (milligram) mg administered once daily for the first week of treatment (titration phase) then 20 mg administered once daily for the next 7 weeks of treatment, followed by placebo capsules administered once daily as appropriate for 1 week (taper/transition phase).
- Desvenlafaxine Succinate Sustained Release (DVS SR): DVS SR capsules 10 or 20 mg (based on weight at the baseline visit) administered once daily for the first week of treatment (titration phase) then 25, 35 or 50 mg (based on weight at the baseline visit) administered once daily for the next 7 weeks of treatment, followed by 10 or 20 mg (based on weight at the baseline visit) (taper phase) or 25 mg (transition phase) administered once daily as appropriate for 1 week.
Period: Overall Study
Arm/Group | Placebo | Fluoxetine | Desvenlafaxine Succinate Sustained Release (DVS SR)
Started | 112 | 113 | 115
Treated | 112 | 112 | 115
Completed | 99 | 99 | 99
Not Completed | 13 | 14 | 16
Not completed — Lack of Efficacy | 3 | 0 | 1
Not completed — Lost to Follow-up | 4 | 5 | 6
Not completed — Protocol Violation | 1 | 0 | 3
Not completed — Withdrawal by Subject | 2 | 7 | 2
Not completed — Other | 1 | 0 | 2
Not completed — Adverse Event | 2 | 1 | 2
Not completed — Randomized but not treated | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Safety population - included all randomized participants who received at least 1 dose of study drug.
Groups:
- Fluoxetine: Fluoxetine capsules 10 mg administered once daily for the first week of treatment (titration phase) then 20 mg administered once daily for the next 7 weeks of treatment, followed by placebo capsules administered once daily for 1 week as appropriate (taper/transition phase).
- DVS SR: DVS SR capsules 10 or 20 mg (based on weight at the baseline visit) administered once daily for the first week of treatment (titration phase) then 25, 35 or 50 mg (based on weight at the baseline visit) administered once daily for the next 7 weeks of treatment, followed by 10 or 20 mg (based on weight at the baseline visit) (taper phase) or 25 mg (transition phase) administered once daily as appropriate for 1 week.
- Total: Total of all reporting groups
Arm/Group | Placebo | Fluoxetine | DVS SR | Total
Number analyzed (Participants) | 112 | 112 | 115 | 339
Age, Continuous [Mean (Standard Deviation); unit: Years] | 12.6 (2.89) | 12.6 (2.89) | 12.9 (3.12) | 12.7 (2.96)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 64 | 57 | 63 | 184
  Male | 48 | 55 | 52 | 155

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline to Week 8 in the Children's Depression Rating Scale, Revised (CDRS-R) Total Score
Description: Clinician-rated interview-based scale (with both child and parent or guardian) to assess 17 distinct symptom areas to derive an index of depression severity. Discrepancies between informants' responses were resolved by using most impaired rating given by valid informant. Rated on a 7-point scale; range from 1 (no impairment) to 7 (indicates greater impairment). Total score calculated as sum of the 17 items (range 1 to 119); higher score indicates greater impairment. Adjusted mean presented.
Time Frame: Baseline and Week 8
Population: Intention-To-Treat (ITT) Population - included all randomized participants who received at least 1 dose of study drug, had a baseline primary efficacy assessment, and had at least one post-baseline primary efficacy assessment.
Measure: Mean (Standard Error); unit: Score on a Scale
Arm/Group | Placebo | Fluoxetine | DVS SR
Number analyzed (Participants) | 99 | 101 | 99
Score on a Scale | -23.07 (1.18) | -24.79 (1.17) | -22.61 (1.17)
Statistical Analysis 1: Comparison: Placebo vs Fluoxetine; Fluoxetine versus Placebo; Test type: Superiority or Other; p = 0.226, Mixed-effects model for repeated measure; Mixed-effects model for repeated measures (MMRM); Mean Difference (Final Values) = 1.71, 95% CI 2-sided [-1.06 to 4.48] — Adjusted mean difference = placebo - fluoxetine
Statistical Analysis 2: Comparison: Placebo vs DVS SR; DVS SR versus Placebo; Test type: Superiority or Other; p = 0.739, MMRM; Mean Difference (Final Values) = -0.47, 95% CI 2-sided [-3.23 to 2.30] — Adjusted mean difference = Placebo - DVS SR

2. Secondary Outcome: Change From Baseline to Week 8 in the Clinical Global Impression of Severity (CGI-S) Score
Description: A 7-point clinician rated scale to assess severity of participant's current illness state; range: 1 (normal - not ill at all) to 7 (among the most extremely ill patients). Higher score = more affected. Change: score at observation minus score at baseline. Adjusted mean presented.
Time Frame: Baseline and Week 8
Population: ITT Population
Measure: Mean (Standard Error); unit: Score on a Scale
Arm/Group | Placebo | Fluoxetine | DVS SR
Number analyzed (Participants) | 99 | 101 | 99
Score on a Scale | -1.71 (0.12) | -1.88 (0.12) | -1.70 (0.11)
Statistical Analysis 1: Comparison: Placebo vs Fluoxetine; Fluoxetine versus Placebo; Test type: Superiority or Other; p = 0.224, MMRM; Mean Difference (Final Values) = 0.18, 95% CI 2-sided [-0.11 to 0.46] — Adjusted mean difference = Placebo - Fluoxetine
Statistical Analysis 2: Comparison: Placebo vs DVS SR; DVS SR versus Placebo; Test type: Superiority or Other; p = 0.944, MMRM; Mean Difference (Final Values) = -0.01, 95% CI 2-sided [-0.29 to 0.27] — Adjusted mean difference = Placebo - DVS SR

3. Secondary Outcome: Percentage of Participants by Clinical Global Impression Improvement (CGI-I) Score at Weeks 1, 2, 3, 4, 6, and 8
Description: A 7-point clinician rated scale ranging from 1 (very much improved) to 7 (very much worse). Improvement is defined as a score of 1 (very much improved), 2 (much improved), or 3 (minimally improved) on the scale. Higher score = more affected.
Time Frame: Baseline and Weeks 1, 2, 3, 4, 6, and 8
Population: ITT Population
Measure: Number; unit: Percentage of Participants
Arm/Group | Placebo | Fluoxetine | DVS SR
Number analyzed (Participants) | 105 | 105 | 111
Percentage of Participants
  Week 1, Very Much Improved (n=102, 101, 111) | 1.0 | 3.0 | 2.7
  Week 1, Much Improved (n=102, 101, 111) | 7.8 | 11.9 | 6.3
  Week 1, Minimally Improved (n=102, 101, 111) | 46.1 | 35.6 | 43.2
  Week 1, No Change (n=102, 101, 111) | 43.1 | 47.5 | 45.9
  Week 1, Minimally Worse (n=102, 101, 111) | 2.0 | 2.0 | 1.8
  Week 1, Much Worse (n=102, 101, 111) | 0 | 0 | 0
  Week 1, Very Much Worse (n=102, 101, 111) | 0 | 0 | 0
  Week 2, Very Much Improved (n=103, 105, 110) | 3.9 | 6.7 | 3.6
  Week 2, Much Improved (n=103, 105, 110) | 25.2 | 26.7 | 31.8
  Week 2, Minimally Improved (n=103, 105, 110) | 38.8 | 42.9 | 44.5
  Week 2, No Change (n=103, 105, 110) | 30.1 | 22.9 | 19.1
  Week 2, Minimally Worse (n=103, 105, 110) | 1.9 | 1.0 | 0.9
  Week 2, Much Worse (n=103, 105, 110) | 0 | 0 | 0
  Week 2, Very Much Worse (n=103, 105, 110) | 0 | 0 | 0
  Week 3, Very Much Improved (n=105, 102, 107) | 13.3 | 14.7 | 7.5
  Week 3, Much Improved (n=105, 102, 107) | 29.5 | 36.3 | 42.1
  Week 3, Minimally Improved (n=105, 102, 107) | 41.0 | 36.3 | 38.3
  Week 3, No Change (n=105, 102, 107) | 15.2 | 11.8 | 11.2
  Week 3, Minimally Worse (n=105, 102, 107) | 1.0 | 1.0 | 0.9
  Week 3, Much Worse (n=105, 102, 107) | 0 | 0 | 0
  Week 3, Very Much Worse (n=105, 102, 107) | 0 | 0 | 0
  Week 4, Very Much Improved (n=101, 101, 100) | 15.8 | 13.9 | 20.0
  Week 4, Much Improved (n=101, 101, 100) | 38.6 | 47.5 | 44.0
  Week 4, Minimally Improved (n=101, 101, 100) | 29.7 | 27.7 | 25.0
  Week 4, No Change (n=101, 101, 100) | 13.9 | 9.9 | 10.0
  Week 4, Minimally Worse (n=101, 101, 100) | 2.0 | 1.0 | 1.0
  Week 4, Much Worse (n=101, 101, 100) | 0 | 0 | 0
  Week 4, Very Much Worse (n=101, 101, 100) | 0 | 0 | 0
  Week 6, Very Much Improved (n=100, 100, 102) | 18.0 | 26.0 | 23.5
  Week 6, Much Improved (n=100, 100, 102) | 41.0 | 45.0 | 45.1
  Week 6, Minimally Improved (n=100, 100, 102) | 34.0 | 24.0 | 20.6
  Week 6, No Change (n=100, 100, 102) | 6.0 | 5.0 | 9.8
  Week 6, Minimally Worse (n=100, 100, 102) | 0 | 0 | 1.0
  Week 6, Much Worse (n=100, 100, 102) | 1.0 | 0 | 0
  Week 6, Very Much Worse (n=100, 100, 102) | 0 | 0 | 0
  Week 8, Very Much Improved (n=99, 101, 99) | 27.3 | 30.7 | 23.2
  Week 8, Much Improved (n=99, 101, 99) | 35.4 | 47.5 | 45.5
  Week 8, Minimally Improved (n=99, 101, 99) | 32.3 | 16.8 | 21.2
  Week 8, No Change (n=99, 101, 99) | 4.0 | 4.0 | 9.1
  Week 8, Minimally Worse (n=99, 101, 99) | 1.0 | 1.0 | 1.0
  Week 8, Much Worse (n=99, 101, 99) | 0 | 0 | 0
  Week 8, Very Much Worse (n=99, 101, 99) | 0 | 0 | 0
Statistical Analysis 1: Comparison: Placebo vs Fluoxetine; Fluoxetine versus Placebo - Week 1; Test type: Superiority or Other; p = 0.924, Cochran-Mantel-Haenszel — P-value obtained from the Cochran-Mantel-Haenszel test for the alternative hypothesis of "Row Mean Scores Differences"
Statistical Analysis 2: Comparison: Placebo vs DVS SR; DVS SR versus Placebo - Week 1; Test type: Superiority or Other; p = 0.698, Cochran-Mantel-Haenszel — P-value obtained from the Cochran-Mantel-Haenszel test for the alternative hypothesis of "Row Mean Scores Differences"
Statistical Analysis 3: Comparison: Placebo vs Fluoxetine; Fluoxetine versus Placebo - Week 2; Test type: Superiority or Other; p = 0.214, Cochran-Mantel-Haenszel — P-value obtained from the Cochran-Mantel-Haenszel test for the alternative hypothesis of "Row Mean Scores Differences"
Statistical Analysis 4: Comparison: Placebo vs DVS SR; DVS SR versus Placebo - Week 2; Test type: Superiority or Other; p = 0.113, Cochran-Mantel-Haenszel — P-value obtained from the Cochran-Mantel-Haenszel test for the alternative hypothesis of "Row Mean Scores Differences"
Statistical Analysis 5: Comparison: Placebo vs Fluoxetine; Fluoxetine versus Placebo - Week 3; Test type: Superiority or Other; p = 0.314, Cochran-Mantel-Haenszel — P-value obtained from the Cochran-Mantel-Haenszel test for the alternative hypothesis of "Row Mean Scores Differences"
Statistical Analysis 6: Comparison: Placebo vs DVS SR; DVS SR versus Placebo - Week 3; Test type: Superiority or Other; p = 0.659, Cochran-Mantel-Haenszel — P-value obtained from the Cochran-Mantel-Haenszel test for the alternative hypothesis of "Row Mean Scores Differences"
Statistical Analysis 7: Comparison: Placebo vs Fluoxetine; Fluoxetine versus Placebo - Week 4; Test type: Superiority or Other; p = 0.577, Cochran-Mantel-Haenszel — P-value obtained from the Cochran-Mantel-Haenszel test for the alternative hypothesis of "Row Mean Scores Differences"
Statistical Analysis 8: Comparison: Placebo vs DVS SR; DVS SR versus Placebo - Week 4; Test type: Superiority or Other; p = 0.187, Cochran-Mantel-Haenszel — P-value obtained from the Cochran-Mantel-Haenszel test for the alternative hypothesis of "Row Mean Scores Differences"
Statistical Analysis 9: Comparison: Placebo vs Fluoxetine; Fluoxetine versus Placebo - Week 6; Test type: Superiority or Other; p = 0.051, Cochran-Mantel-Haenszel — P-value obtained from the Cochran-Mantel-Haenszel test for the alternative hypothesis of "Row Mean Scores Differences"
Statistical Analysis 10: Comparison: Placebo vs DVS SR; DVS SR versus Placebo - Week 6; Test type: Superiority or Other; p = 0.266, Cochran-Mantel-Haenszel — P-value obtained from the Cochran-Mantel-Haenszel test for the alternative hypothesis of "Row Mean Scores Differences"
Statistical Analysis 11: Comparison: Placebo vs Fluoxetine; Fluoxetine versus Placebo - Week 8; Test type: Superiority or Other; p = 0.095, Cochran-Mantel-Haenszel — P-value obtained from the Cochran-Mantel-Haenszel test for the alternative hypothesis of "Row Mean Scores Differences"
Statistical Analysis 12: Comparison: Placebo vs DVS SR; DVS SR versus Placebo - Week 8; Test type: Superiority or Other; p = 0.852, Cochran-Mantel-Haenszel — P-value obtained from the Cochran-Mantel-Haenszel test for the alternative hypothesis of "Row Mean Scores Differences"

4. Secondary Outcome: Percentage of Participants With a CGI-I Response Defined as a Score of 'Very Much Improved' or 'Much Improved'
Description: as for outcome 3
Time Frame: Weeks 1, 2, 3, 4, 6, and 8
Population: ITT Population
Measure: Number; unit: Percentage of Participants
Arm/Group | Placebo | Fluoxetine | DVS SR
Number analyzed (Participants) | 105 | 105 | 111
Percentage of Participants
  Week 1 (n=102, 101, 111) | 8.82 | 14.85 | 9.01
  Week 2 (n=103, 105, 110) | 29.13 | 33.33 | 35.45
  Week 3 (n=105, 102, 107) | 42.86 | 50.98 | 49.53
  Week 4 (n=101, 101, 100) | 54.46 | 61.39 | 64.00
  Week 6 (n=100, 100, 102) | 59.00 | 71.00 | 68.63
  Week 8 (n=99, 101, 99) | 62.63 | 78.22 | 68.69
Statistical Analysis 1: Comparison: Placebo vs Fluoxetine; Fluoxetine versus Placebo - Week 1; Test type: Superiority or Other; p = 0.186, Regression, Logistic; Odds Ratio (OR) = 0.550, 95% CI 2-sided [0.226 to 1.335] — Logistic Regression using Response (Y/N) at each time point (excluding Week 9) as a response variable and treatment, age group and country as factors
Statistical Analysis 2: Comparison: Placebo vs DVS SR; DVS SR versus Placebo - Week 1; Test type: Superiority or Other; p = 0.984, Regression, Logistic; Odds Ratio (OR) = 0.990, 95% CI 2-sided [0.382 to 2.567] — [estimate comment as in outcome 4, analysis 1]
Statistical Analysis 3: Comparison: Placebo vs Fluoxetine; Fluoxetine versus Placebo - Week 2; Test type: Superiority or Other; p = 0.462, Regression, Logistic; Odds Ratio (OR) = 0.795, 95% CI 2-sided [0.431 to 1.465] — [estimate comment as in outcome 4, analysis 1]
Statistical Analysis 4: Comparison: Placebo vs DVS SR; DVS SR versus Placebo - Week 2; Test type: Superiority or Other; p = 0.297, Regression, Logistic; Odds Ratio (OR) = 0.726, 95% CI 2-sided [0.399 to 1.324] — [estimate comment as in outcome 4, analysis 1]
Statistical Analysis 5: Comparison: Placebo vs Fluoxetine; Fluoxetine versus Placebo - Week 3; Test type: Superiority or Other; p = 0.194, Regression, Logistic; Odds Ratio (OR) = 0.688, 95% CI 2-sided [0.391 to 1.210] — [estimate comment as in outcome 4, analysis 1]
Statistical Analysis 6: Comparison: Placebo vs DVS SR; DVS SR versus Placebo - Week 3; Test type: Superiority or Other; p = 0.272, Regression, Logistic; Odds Ratio (OR) = 0.732, 95% CI 2-sided [0.419 to 1.277] — [estimate comment as in outcome 4, analysis 1]
Statistical Analysis 7: Comparison: Placebo vs Fluoxetine; Flouxetine versus Placebo - Week 4; Test type: Superiority or Other; p = 0.313, Regression, Logistic; Odds Ratio (OR) = 0.748, 95% CI 2-sided [0.426 to 1.314] — [estimate comment as in outcome 4, analysis 1]
Statistical Analysis 8: Comparison: Placebo vs DVS SR; DVS SR versus Placebo - Week 4; Test type: Superiority or Other; p = 0.157, Regression, Logistic; Odds Ratio (OR) = 0.663, 95% CI 2-sided [0.376 to 1.171] — [estimate comment as in outcome 4, analysis 1]
Statistical Analysis 9: Comparison: Placebo vs Fluoxetine; Flouxetine versus Placebo - Week 6; Test type: Superiority or Other; p = 0.072, Regression, Logistic; Odds Ratio (OR) = 0.579, 95% CI 2-sided [0.319 to 1.050] — [estimate comment as in outcome 4, analysis 1]
Statistical Analysis 10: Comparison: Placebo vs DVS SR; DVS SR versus Placebo - Week 6; Test type: Superiority or Other; p = 0.135, Regression, Logistic; Odds Ratio (OR) = 0.640, 95% CI 2-sided [0.356 to 1.149] — [estimate comment as in outcome 4, analysis 1]
Statistical Analysis 11: Comparison: Placebo vs Fluoxetine; Flouxetine versus Placebo - Week 8; Test type: Superiority or Other; p = 0.017, Regression, Logistic; Odds Ratio (OR) = 0.465, 95% CI 2-sided [0.249 to 0.871] — [estimate comment as in outcome 4, analysis 1]
Statistical Analysis 12: Comparison: Placebo vs DVS SR; DVS SR versus Placebo - Week 8; Test type: Superiority or Other; p = 0.343, Regression, Logistic; Odds Ratio (OR) = 0.751, 95% CI 2-sided [0.415 to 1.357] — [estimate comment as in outcome 4, analysis 1]

ADVERSE EVENTS:
Time Frame: Adverse events (AEs) were recorded from informed consent and assent through the first follow up visit (Week 11) for non-serious AEs; the second follow up visit (Week 13) for serious AEs (SAEs); or at Week 9 for participants entering the extension study.
Description: The same event may appear as both an AE and an SAE. However, what is presented are distinct events. An event may be categorized as serious in 1 participant and as non-serious in another participant, or 1 participant may have experienced both a serious and non-serious event during the study.
Arm/Group | Placebo | Fluoxetine | DVS SR
Serious Adverse Events (participants affected / at risk) | 0/112 | 2/112 | 2/115
Other Adverse Events (participants affected / at risk) | 44/112 | 39/112 | 47/115
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=112) | Fluoxetine (N=112) | DVS SR (N=115)
Disinhibition (Psychiatric disorders) | 0 | 0 | 1
Suicidal ideation (Psychiatric disorders) | 0 | 1 | 1
Suicide attempt (Psychiatric disorders) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=112) | Fluoxetine (N=112) | DVS SR (N=115)
Abdominal pain upper (Gastrointestinal disorders) | 7 | 9 | 15
Nausea (Gastrointestinal disorders) | 10 | 13 | 8
Vomiting (Gastrointestinal disorders) | 4 | 7 | 5
Fatigue (General disorders) | 2 | 6 | 2
Influenza (Infections and infestations) | 0 | 2 | 6
Nasopharyngitis (Infections and infestations) | 8 | 7 | 6
Upper respiratory tract infection (Infections and infestations) | 6 | 4 | 6
Dizziness (Nervous system disorders) | 6 | 3 | 7
Headache (Nervous system disorders) | 21 | 16 | 19

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less